CLINICAL TRIAL: NCT06722898
Title: Rapid Blood Alcohol Concentration Reduction with Nutraceutical Blend Study
Brief Title: Rapid BAC Reduction with Nutraceutical Blend Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical Life Care Planners, LLC (Other)
Responsible Party: Principal Investigator, Gregory L Smith, MD, MPH, Primary Investigator, Medical Life Care Planners, LLC
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 000011
Record Dates: First submitted 2024-10-31; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Alcohol Consumption; Alcohol; Hangover Symptoms, NAC; Veisalgia
Keywords: alcohol; blood alcohol; alcohol intoxication; alcohol impairment; BAC; BAC reduction; alcohol half-life; blood alcohol concentration; veisalgia; hangover
MeSH Terms: conditions — Alcohol Drinking; Alcoholic Intoxication | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Liquid (Active Comparator)
  Interventions: Dietary Supplement: Supplement

INTERVENTIONS:
Dietary Supplement: Supplement — Contains ingredients believed to reduce Blood Alcohol Concentration and symptoms of alcohol impairment.
  Arms: Liquid
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Study Title: Nutritional Supplement to Rapidly Decrease Blood Alcohol Concentration (BAC): Safety and Efficacy Study Design: Double-blind, randomized, placebo-controlled clinical trial Objective: Evaluate safety and efficacy of a nutritional supplement to rapidly decrease blood alcohol concentration (BAC), alcohol-induced impairment, and hangover symptoms after excessive alcohol consumption.

Primary Outcomes:

BAC reduction rate/extent (BACtrack S80™ breathalyzer) Cognitive/physical impairment change (DRUID app™)

Secondary Outcome:

Hangover symptom reduction (Acute Hangover Scale) Participants: 35 participants, recruited via social media Duration: 2 weeks, 2 testing sessions (4 hours each) Location: Closed facility in St. Petersburg, FL

Procedure:

Subjects consume standardized alcohol (1g ethanol/kg body weight) 40-minute drinking period BAC and impairment measurements Administration of test formulation or placebo

Measurements:

BAC: Baseline, 40min, 15min, 30min, 60min, 90min post-drinking Impairment: Baseline, 15min, 30min, 60min post-drinking Hangover: Next morning via text message

Safety Measures:

GRAS ingredients Lab testing of formulations Medical screening Adverse effect questionnaires Pregnancy tests BAC &lt;0.08% before leaving

Key Features:

Paired measurements: active vs. placebo for mini-drink and capsule formulations Uber transportation provided Strict inclusion/exclusion criteria

Data Analysis:

Electronic data entry Blinded submission for statistical analysis Paired comparisons and multiple statistical tests

This study aims to provide robust data on the efficacy in mitigating alcohol's effects, potentially offering a new tool for reducing alcohol-related impairment and hangover symptoms. The design prioritizes safety, consistency, and scientific rigor to ensure reliable results.

DETAILED DESCRIPTION:
Study Title: Nutraceutical Safety and Efficacy Study

Introduction:

The nutraceutical Safety and Efficacy Study is a comprehensive clinical trial designed to evaluate a novel formulation aimed at rapidly decreasing blood alcohol concentration (BAC), alcohol-induced impairment, and veisalgia (hangover) symptoms following excessive alcohol consumption. This study addresses a significant public health concern by potentially offering a method to mitigate the negative effects of alcohol overconsumption.

Study Design:

This is a triple-blinded, randomized, placebo-controlled clinical trial. The triple-blind nature ensures that the subjects, investigators, and data analysts are unaware of the treatment assignments, minimizing bias in the results.

Primary Objectives:

To determine the rate and extent of BAC reduction after administration of nutraceutical compared to placebo.

To assess the change in cognitive and physical impairment due to nutraceutical supplement after excessive alcohol consumption.

Secondary Objective:

To evaluate the reduction in hangover symptoms the morning after excessive alcohol consumption when active compared to placebo.

Study Population:

The study will recruit 70 subjects (35 per arm) from the Tampa Bay area through social media. Key inclusion criteria include:

Age 21 or older Regular social alcohol use Not naive to consuming more than 4 drinks at once Ability to attend all three sessions Ownership of a smartphone with texting capabilities

Exclusion criteria encompass:

Alcohol Use Disorder (AUDIT score ≥8) Use of certain medications (e.g., Antabuse, beta-lactam antibiotics) Current use of psychoactive products or illegal substances Active medical conditions precluding excessive alcohol use Pregnancy or unknown pregnancy status Current involvement in the criminal justice system

Study Duration and Timeline:

The study will span 4 weeks, with three testing sessions scheduled on Sundays: August 15th, August 22nd, and October 5th, 2024. Each session will last approximately 4 hours, from 4 PM to 8 PM. The final statistical analysis and preparation for journal submission are expected to be completed by early November 2024.

Study Location:

All sessions will be conducted at a centrally located closed bar in St. Petersburg, FL, ensuring a controlled environment for the study.

Intervention:

The study will test two formulations:

Capsule form Mini-drink form

Each formulation will be compared against a matching placebo. The active ingredients and placebos will be provided. The exact composition is proprietary, but it consists of Generally Recognized as Safe (GRAS) ingredients.

Study Procedure:

Each subject will participate in three sessions, receiving either the active formulation or placebo in a randomized order. The procedure for each session is as follows:

Subjects arrive and consume a standardized meal (one slice of pizza or equivalent).

Baseline measurements are taken (BAC and impairment tests). Subjects consume a 20 oz container of vodka and flavoring (1g ethanol per kg of body weight) over a 40-minute period.

Immediately after drinking, BAC is measured, and impairment tests are conducted.

Subjects receive either the active formulation or placebo. BAC measurements are taken at 15, 30, 60, and 90 minutes post-drinking. Impairment tests are conducted at 15, 30, and 60 minutes post-drinking. Subjects remain at the facility until their BAC is below 0.08%, then are provided Uber transportation home.

The following morning at 8 AM, subjects complete a hangover questionnaire via text message.

Outcome Measures:

Blood Alcohol Concentration (BAC):

Instrument: BACtrack S80™ breathalyzer (US FDA 510(k) approved) Measurement points: Baseline, immediately after drinking (40 minutes), then at 15, 30, 60, and 90 minutes post-drinking Analysis: Rate and extent of BAC reduction compared to placebo

Cognitive and Physical Impairment:

Primary instrument: DRUID app™

Secondary measures:

1. Horizontal Gaze Nystagmus (HGN) test
2. One-leg Stand test
3. Computer-assisted testing for reaction time, sustained attention, and decision making (www.HumanBenchMark.com) Measurement points: Baseline, 15, 30, and 60 minutes post-drinking Analysis: Change in impairment scores compared to placebo

Hangover Symptoms:

Instrument: Acute Hangover Scale (AHS™) Description: 9-question survey, rating symptoms on a scale of 0-7 Administration: Via text message at 8 AM the morning after each session Analysis: Comparison of hangover symptom scores between and placebo conditions

Safety Measures:

Use of GRAS ingredients in formulations Independent lab testing and certificate of analysis for all test formulations Thorough medical screening of subjects Administration of standardized adverse effect questionnaires Urine pregnancy tests for women of childbearing age before each session Ensuring subjects' BAC is below 0.08% before leaving the facility Provision of Uber transportation to and from each session

Subject Consistency and Compliance:

To ensure physiological similarity across sessions, subjects will:

Drink a quart of water starting 4 hours before each session Refrain from eating or drinking (except water) for 4 hours before each session Consume the same standardized meal at the beginning of each session Agree to abstain from alcohol and euphoric substances for 24 hours after each session

Staffing:

A minimum of 14 support staff will be on-site to ensure efficient flow of subjects through each session. Dr. Gregory L. Smith and a medical assistant will conduct the physical impairment testing throughout the study sessions.

Data Collection and Management:

Data will be collected via a pre-prepared electronic data entry system for each individual subject. All data will be blinded and submitted electronically for separate statistical analysis.

Statistical Analysis:

The study will employ separate statistical analyses for paired comparisons of the capsule formulation and the mini-drink formulation. Multiple statistical tests will be conducted to determine statistical significance within the paired data, separately for each formulation and as combined data. The study aims for 80% statistical power with a p-value 0.05.

Ethical Considerations:

Institutional Review Board (IRB) approval will be obtained from the Medical Life Care Planners IRB.

The study will be registered on ClinicalTrials.gov and assigned a National Clinical Trial (NCT) number.

Informed consent will be obtained from all participants prior to study enrollment.

Subjects' privacy and data confidentiality will be maintained throughout the study.

Potential Impact:

If proven effective, could have significant implications for public health and safety. It could potentially:

Reduce the risk of alcohol-related accidents and injuries Mitigate productivity losses due to hangovers Provide a tool for responsible alcohol consumption

However, it's crucial to note that the product should not be seen as a means to enable excessive drinking or as a substitute for responsible alcohol consumption.

Limitations:

Single-center study, which may limit generalizability Relatively short duration of follow-up (next morning only) Potential for recall bias in self-reported hangover symptoms Unable to control for all factors that might influence alcohol metabolism or hangover severity (e.g., genetics, overall health status)

Future Directions:

Depending on the results of this initial study, future research could explore:

Long-term safety and efficacy Effects on different populations (e.g., varying age groups, ethnicities) Potential interactions with medications or medical conditions Optimal dosing and timing of administration Physiological mechanisms of action

Conclusion:

The Nutraceutical Safety and Efficacy Study represents a rigorous approach to evaluating a novel intervention for mitigating the effects of alcohol overconsumption. By employing a triple-blind, randomized, placebo-controlled design with multiple outcome measures, this study aims to provide robust evidence regarding the safety and efficacy. The results could have significant implications for public health strategies related to alcohol consumption and its associated risks.

ELIGIBILITY:
Inclusion Criteria:

* Over age 21
* Provide signed Informed Consent form electronically in advance of the first study date.
* Provided signed Acknowledgement Form of what is required as part of the study, including use of Uber for transportation to and from each session.
* Not taking certain prescription medications to be listed.
* No history of alcohol or substance abuse issues or alcohol-related medical conditions.
* No history of liver disease.
* No history of significant violent behavior.
* Uses alcohol socially on a regular basis.
* Not naïve to consuming more than 4 drinks at one time.
* Not pregnant or at risk for being pregnant.
* Able to attend all three session dates.
* Own smartphone with text messaging abilities.

Exclusion Criteria:

* Score consistent with Alcohol Use Disorder on the Alcohol Use Disorder Identification Test (AUDIT) a 10 question self-report tool developed by the World Health Organization (WHO).
* Ongoing or regular use of any of the following medications for medical conditions: Antabuse (disulfiram): (Slows alcohol metabolism by inhibiting the elimination of acetaldehyde), Beta-lactam antibiotics: (Some, such as cefmandole, cefoperazone, and moxalactam, can cause a disulfiram-like reaction when alcohol is consumed), Nitrates (Can cause a disulfiram-like reaction when alcohol is consumed), Sulfonylureas (Longer acting ones, such as chlorpropamide and tolbutamide, can cause a disulfiram-like reaction when alcohol is consumed, as well as Pyrazoles and isobutyramide, Inhibit ADH, which decreases the rate at which alcohol is eliminated.)
* Current use of medications likely to be synergistic with one-time excessive use of alcohol: opioids, benzodiazepines, anti-histamines.
* Current use of psychoactive products such as delta 8 or delta 9 tetrahydrocannabinol (THC), Kava, Kratom or psychedelic mushroom (psilocybin).
* Current use of any illegal drug or substance, that includes, but is not limited to -cocaine, methamphetamine, MDMA (ecstasy, molly).
* Active medical conditions that would preclude one-time excessive use of alcohol: Liver disease, diabetes mellitus, seizure disorder/epilepsy, uncontrolled hypertension, cardiac arrhythmia, Multiple Sclerosis, Schizophrenia, Traumatic Brain Injury (TBI), active peptic ulcer disease (PUD), and opioid use disorder

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-07 (Estimated)

PRIMARY OUTCOMES:
Blood Alcohol Concentration | 90 minutes
  The first primary outcome measure will be the rate and extent of Blood Alcohol Concentration (BAC) reduction due to the effects of administering BAC Down™ after excessive consumption of alcohol, tested using a BACtrack S80™ (US FDA 501(k)) advanced technology breathalyzer.
Alcohol Impairment | 90 minutes
  The second primary outcome measure will be change in cognitive/physical impairment due to the effects of administering BAC Down™ after excessive alcohol consumption. The DRUID app™ will be used to measure cognitive and motor impairment. Each subject will have a standard training session with the use of the DRUID app on their phone.

SECONDARY OUTCOMES:
Reduction of Hangover Symptoms | 12-24 hours after study completion
  The secondary outcome measure is subjective reduction in veisalgia (hangover) symptoms using a standardized self-reported questionnaire the morning after excessive alcohol consumption in combination with BAC Down™ or placebo, utilizing The Acute Hangover Scale (AHS™), a 9-question survey where each symptom is rated on a scale for 0-7. Each subject will be provided with the AHS™ questionnaire via a text the morning following the three test dates. The text will be sent at the expected "awakening time" according to the subject to facilitate consistency and validity.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory L Smith, MD, MPH, Principal Investigator — NeX Therapeutics
Locations (1):
- The Warehouse St. Pete, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected data points without any personal identifying information.
Supporting Information: Study Protocol, ICF
Time Frame: 1 year